CLINICAL TRIAL: NCT01571388
Title: A Phase 1 Study To Evaluate The Single Dose Pharmacokinetics Of Dacomitinib (PF-00299804) In Subjects With Impaired Hepatic Function
Brief Title: A Study To Compare Pharmacokinetics Of Dacomitinib (PF-00299804) Between Healthy Subjects And Subjects With Mild And Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A7471018
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Healthy; Otherwise Healthy Volunteers With Mild or Moderate Hepatic Dysfunction
Keywords: dacomitinib; PF-00299804; hepatic impairment; pharmacokinetics
MeSH Terms: interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Healthy Subjects to receive dacomitinib
  Interventions: Drug: dacomitinib
- Group 2 (Experimental): Subjects with mildly impaired hepatic function to receive dacomitinib
  Interventions: Drug: dacomitinib
- Group 3 (Experimental): Subjects with moderately impaired hepatic function to receive dacomitinib
  Interventions: Drug: dacomitinib

INTERVENTIONS:
Drug: dacomitinib — Subjects to receive 30 mg tablets of dacomitinib on Day 1 of Period 1.
  Arms: Group 1
Drug: dacomitinib — Subjects to receive 30 mg tablets of dacomitinib on Day 1 of Period 1.
  Arms: Group 2
Drug: dacomitinib — Subjects to receive 30 mg tablets of dacomitinib on Day 1 of Period 1.
  Arms: Group 3

SUMMARY:
The study will determine if there are differences in how dacomitinib is absorbed and eliminated between healthy subjects and subjects with mild and moderately impaired hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 years of age to <75 years of age. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests. Liver function tests, albumin and prothrombin time must be within normal range.
* Body Mass Index (BMI) of 18 to 35 kg/m2;
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Subjects in the normal hepatic function group (Group 1): No known or suspected hepatic impairment.
* For subjects in the hepatic impairment groups (Groups 2 and 3):

  * Should satisfy the criteria for Class A or B of the modified Child-Pugh classification
  * A diagnosis of hepatic dysfunction due to hepatocellular disease (and not secondary to any acute ongoing hepatocellular process) documented by medical history, physical examination, liver biopsy, hepatic ultrasound, CT scan, or MRI.
  * Stable hepatic impairment, defined as no clinically significant change in disease status within the last 30 days, as documented by the subject's recent medical history
  * Must be on a stable dose of medication and/or treatment regimen.

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy, chronic diarrhea, rapid transit).
* A positive urine drug screen.
* Females of childbearing potential, including those with tubal ligation. [To be considered for enrollment, women of at least 45 years of age who are postmenopausal (defined as being amenorrheic for at least 2 years) must have confirmatory FSH test results at screening].
* In addition, subjects in the hepatic impairment groups (Groups 2 and 3) presenting with any of the following will not be included in the trial:

  * Hepatic carcinoma and hepatorenal syndrome or life expectancy <1 year.
  * Undergone porta-caval shunt surgery.
  * History of gastrointestinal hemorrhage due to esophageal varices or peptic ulcers less than one month prior to study entry.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 2 weeks
  Maximal plasma concentration (Cmax) for dacomitinib
Plasma area under plasma concentration-time curve from time zero to time infinity post dose (AUCinf) for dacomitinib | 2 weeks

SECONDARY OUTCOMES:
Area under the Concentration-Time Curve (AUC);Plasma area under plasma concentration-time curve from time zero to 24 hours post dose (AUC24) for dacomitinib | 2 weeks
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Plasma area under plasma concentration-time curve from time zero to 216 hours post dose (AUC216) for dacomitinib | 2 weeks
Plasma area under plasma concentration-time curve from time zero to time of last quantifiable concentration post dose (AUClast) for dacomitinib | 2 weeks
Time of first observed maximal plasma concentration (Tmax) for dacomitinib | 2 weeks
Plasma elimination half life (t1/2) of dacomitinib | 2 weeks
Apparent plasma clearance (CL/F) of dacomitinib | 2 weeks
Apparent volume of distribution (Vz/F) of dacomitinib | 2 weeks
Fraction of unbound dacomitinib in plasma (fu) | 2 weeks
Unbound apparent plasma clearance (CL/F) of dacomitinib , | 2 weeks
Unbound apparent volume of distribution (Vz/F) of dacomitinib | 2 weeks
Unbound Plasma area under plasma concentration-time curve from time zero to time infinity post dose (AUCinf) for dacomitinib | 2 weeks
Unbound plasma area under plasma concentration-time curve from time zero to 24 hours post dose (AUC24) for dacomitinib | 2 weeks
Unbound plasma area under plasma concentration-time curve from time zero to 216 hours post dose (AUC216) for dacomitinib | 2 weeks
Unbound plasma area under plasma concentration-time curve from time zero to time of last quantifiable concentration post dose (AUClast) for dacomitinib | 2 weeks
Maximal unbound plasma concentration (Cmax) for dacomitinib | 2 weeks
Plasma area under plasma concentration-time curve from time zero to time infinity post dose (AUCinf) for PF-05199265 | 2 weeks
Plasma area under plasma concentration-time curve from time zero to 24 hours post dose (AUC24) for PF-05199265 | 2 weeks
Plasma area under plasma concentration-time curve from time zero to 216 hours post dose (AUC216) for PF-05199265 | 2 weeks
Plasma area under plasma concentration-time curve from time zero to time of last quantifiable concentration post dose (AUClast) for PF-05199265 | 2 weeks
Maximal plasma concentration (Cmax) for PF-05199265 | 2 weeks
Time of first observed maximal plasma concentration (Tmax) for PF-05199265 | 2 weeks
Metabolite ratio for plasma area under plasma concentration-time curve from time zero to time infinity post dose (MRAUCinf) | 2 weeks
Metabolite ratio for plasma area under plasma concentration-time curve from time zero to time of last quantifiable concentration post dose (MRAUClast) | 2 weeks
Metabolite ratio for maximal plasma concentration (MRCmax) | 2 weeks
Fraction of unbound PF-05199265 in plasma (fu) | 2 weeks
Unbound plasma area under plasma concentration-time curve from time zero to 24 hours post dose (AUC24) for PF-05199265 | 2 weeks
Unbound plasma area under plasma concentration-time curve from time zero to 216 hours post dose (AUC216) for PF-05199265 | 2 weeks
Unbound plasma area under plasma concentration-time curve from time zero to time of last quantifiable concentration post dose (AUClast) for PF-05199265 | 2 weeks
Unbound Plasma area under plasma concentration-time curve from time zero to time infinity post dose (AUCinf) for PF-05199265 | 2 weeks
Maximal unbound plasma concentration (Cmax) for PF-05199265 | 2 weeks
Overall safety profile as characterized by laboratory abnormalities, observed physical examination, vital signs, ECGs, and adverse event monitoring. | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, South Miami, Florida

REFERENCES:
- [Derived] Piscitelli J, Chen J, LaBadie RR, Salageanu J, Chung CH, Tan W. The Effect of Hepatic Impairment on the Pharmacokinetics of Dacomitinib. Clin Drug Investig. 2022 Mar;42(3):221-235. doi: 10.1007/s40261-022-01125-x. Epub 2022 Feb 23. PMID 35195881
- [Derived] Giri N, Masters JC, Plotka A, Liang Y, Boutros T, Pardo P, O'Connell J, Bello C. Investigation of the impact of hepatic impairment on the pharmacokinetics of dacomitinib. Invest New Drugs. 2015 Aug;33(4):931-41. doi: 10.1007/s10637-015-0256-0. Epub 2015 Jun 6. PMID 26048096
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471018&StudyName=A%20Study%20To%20Compare%20Pharmacokinetics%20Of%20Dacomitinib%20%28PF-00299804%29%20Between%20Healthy%20Subjects%20And%20Subjects%20With%20Mild%20And%20Moderate%20Hepatic%20